CLINICAL TRIAL: NCT01802619
Title: Prevention of Renal Failure by Nitric Oxide in Prolonged Cardiopulmonary Bypass: A Double Blind Randomized Controlled Trial.
Brief Title: Prevention of Renal Failure by Nitric Oxide in Prolonged Cardiopulmonary Bypass.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, chonglei, M.D.& Ph.D., Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20121025-8; 81000232 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2013-02-25; First posted 2013-03-01 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Heart Valve Diseases; Heart; Complications, Valve, Prosthesis; Cardiac Valve Replacement Complication
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- inhaled nitrogen (Placebo Comparator): Using an Inovent (Ikaria Inc, N.J., USA) or volumetrically-calibrated flowmeters, pure nitrogen (placebo) is mixed with pure O2 or air. During CPB the gas mixture is delivered through the extracorporeal oxygenator, after CPB the NO is delivered through the inspiratory limb of the anesthetic or ventilator circuit.
  Interventions: Other: inhaled Nitrogen
- inhaled nitric oxide (Experimental): Using an Inovent (Ikaria Inc, N.J., USA) or volumetrically-calibrated flowmeters, 800 ppm NO gas is mixed with pure O2 or air to obtain a final concentration of 80 ppm NO. During CPB the gas mixture is delivered through the extracorporeal oxygenator, after CPB the gas is delivered through the inspiratory limb of the anesthetic or ventilator circuit. NO, NO2 and O2 and methemoglobin levels are monitored by an unblinded observer.
  Interventions: Other: inhaled nitric oxide

INTERVENTIONS:
Other: inhaled nitric oxide — Nitric oxide administration will commence at the onset of CPB and last for 24 hours. At the end of 24 hours, inhaled NO will be weaned and discontinued while carefully monitoring hemodynamics for a period of 2-4 hours.
  Arms: inhaled nitric oxide
Other: inhaled Nitrogen — Standard gas including nitrogen (the vehicle of the Nitric oxide) administration will commence at the onset of CPB and last for 24 hours. At the end of 24 hours, inhaled gases will be weaned and discontinued while carefully monitoring hemodynamics for a period of 2-4 hours.
  Arms: inhaled nitrogen

SUMMARY:
Prolonged periods of cardiopulmonary bypass (CPB) cause high levels of plasma free haemoglobin(Hb) and are associated with increased morbidity. We hypothesized that repletion of nitric oxide (NO) during and after the surgical procedure on CPB may protect against endothelium dysfunction and organ failure caused by plasma-Hb induced NO scavenging.

DETAILED DESCRIPTION:
Prolonged periods of cardiopulmonary bypass (CPB) cause high levels of plasma free haemoglobin(Hb) and are associated with increased morbidity. We hypothesized that repletion of nitric oxide (NO) during and after the surgical procedure on CPB may protect against endothelium dysfunction and organ failure caused by plasma-Hb induced NO scavenging. There are three possible beneficial mechanisms of delivering NO:

1. Nitric oxide reduces ischemia-reperfusion injury (such as in acute myocardial infarction, stroke, and acute tubular necrosis).
2. Nitric oxide has anti-inflammatory properties. As antioxidants, exogenous NO may reduce injury by counteracting the cytotoxic effects of reactive oxygen species, modulating leukocyte recruitment, edema formation and tissue disruption.
3. Exogenous nitric oxide prevents noxious effects of hemolysis-associated NO dysregulation. During hemolysis, nitric oxide gas oxidized of plasma oxyhemoglobin to methemoglobin, thereby inhibiting endogenous endothelium NO scavenging by cell-free Hb.

NO depletion during hemolysis and its sequelae. The release of plasma free Hb (with Fe2+ iron) by hemolysis avidly scavenges nitric oxide (NO) by the dioxygenation reaction. Elevated plasma ferrous Hb levels can induce a "NO deficiency" state. Reduced vascular nitric oxide levels can contribute to vasoconstriction, inflammation, and thrombosis, potentially contributing to systemic endothelial dysfunction after cardiac surgery with CPB.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Are > 18 years of age
* Elective cardiac or aortic surgery with CPB, when the surgeon plans double valve replacement.
* Stable pre-operative renal function, without dialysis.

Exclusion Criteria:

* Emergent cardiac surgery
* Life expectancy < 1 year
* Hemodynamic instability as defined by a systolic blood pressure <90 mmHg
* Administration of ≥1 Packed Red Blood Cell transfusion in the week before surgery
* X-ray contrast infusion less than 1 week before surgery
* Anticipate administration of nephrotoxic agents, such as hydroxyethyl starch
* Evidence of intravascular or extravascular hemolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
acute kidney injury | an increase of serum creatinine by 50% within 7 days after surgery, or an increase of serum creatinine by 0.3 mg/dl within 2 days after surgery
  acute kidney injury was defined by the KDIGO criteria

SECONDARY OUTCOMES:
Chronic kidney disease | at 30 days, 90 days, and 1 year following ICU admission
  defined as eGFR<60 mL/min/1.73m2
Loss of 25% of eGFR compared to baseline | at 30 days, 90 days, and 1 year following ICU admission
  Loss of 25% of eGFR compared to baseline
Major adverse kidney events (MAKE) | at 30 days, 90 days, and 1 year following ICU admission
  a composite outcome of loss of 25% of eGFR from baseline, end stage renal disease requiring a continuous renal replacement therapy and mortality.
Renal Replacement Therapy | at 30 days, 90 days, and 1 year following ICU admission
  the incidence of need for Renal Replacement Therapy
Incidence of nonfatal stroke and nonfatal myocardial infarction. | at 30 days, 90 days, and 1 year following ICU admission
  Nonfatal stroke will be assessed by the NIH Stroke Scale at baseline before surgery and at 28 days, 60 days, 90 days and 1 year after surgery.
  Nonfatal myocardial infarction is defined by the third universal definition of MI released in 2012 by the ESC/ACCF/AHA/WHF.
Quality of life | at 30 days, 90 days, and 1 year following ICU admission
  The quality of life will be evaluated by the Katz Index of In dependence in Activities of Daily living
overall mortality | at 30 days, 90 days, and 1 year following ICU admission
  all cause mortality

OTHER OUTCOMES:
In-hospital stay | Normally within 30 days, when patients was discharged from ICU
  It is the length of hospital stay
ICU-stay | Normally within 30 days, when patients was discharged from ICU
  It is the length of stay in ICU
Incidence of prolonged ventilation | During hospital stay, normally within 30 days
  Prolonged ventilation is defined as patients remaining on the ventilator for more than 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: lize Xiong, M.D.,Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Hu J, Rezoagli E, Zadek F, Bittner EA, Lei C, Berra L. Free Hemoglobin Ratio as a Novel Biomarker of Acute Kidney Injury After On-Pump Cardiac Surgery: Secondary Analysis of a Randomized Controlled Trial. Anesth Analg. 2021 Jun 1;132(6):1548-1558. doi: 10.1213/ANE.0000000000005381. PMID 33481401
- [Derived] Lei C, Berra L, Rezoagli E, Yu B, Dong H, Yu S, Hou L, Chen M, Chen W, Wang H, Zheng Q, Shen J, Jin Z, Chen T, Zhao R, Christie E, Sabbisetti VS, Nordio F, Bonventre JV, Xiong L, Zapol WM. Nitric Oxide Decreases Acute Kidney Injury and Stage 3 Chronic Kidney Disease after Cardiac Surgery. Am J Respir Crit Care Med. 2018 Nov 15;198(10):1279-1287. doi: 10.1164/rccm.201710-2150OC. PMID 29932345